CLINICAL TRIAL: NCT05678686
Title: Investigation of The Effects of Different Exercise Methods on Swallowing Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Esra Nur ÖZCAN, Lecturer, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMU-EOZCAN-001
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Stroke; Dysphagia; Swallowing Disorder
Keywords: Dysphagia; Stroke; PNF Exercise; CTAR Exercise; Swallowing Rehabilitation
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The physicians who will evaluate imaging methods will not know which arm they are in. In addition patricipants will not know which arm they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine Exercise Group (Active Comparator): Conventional swallowing therapy exercises will be given to the routine exercise group.
  Interventions: Other: Active Comparator: Routine Exercise Group
- PNF Exercise (Experimental): Head-neck PNF (Proprioceptive Neuromuscular Facilitation) movement patterns will be applied to the participants with the combined isometric contraction technique.
  Interventions: Other: Experimental: PNF Exercise
- CTAR Exercise (Experimental): CTAR (Chin Tuck Against Resistance) exercises will be applied to the participants.
  Interventions: Other: Experimental: CTAR Exercise

INTERVENTIONS:
Other: Active Comparator: Routine Exercise Group — Exercises (tongue-palate exercises, tongue base exercises, Masako Maneuver, Mendelson Maneuver, Effortful Swallowing, Supraglottic exercises, thermal tactile stimulation) will be performed 2 days a week for 8 weeks, in total 16 sessions and these exercises applied by the physiotherapist.
  Arms: Routine Exercise Group
Other: Experimental: PNF Exercise — In addition to the practices in the control group, head-neck PNF(Proprioceptive Neuromuscular Facilitation) movement patterns will be applied to both movement patterns by the physiotherapist using the combined isotonic contraction technique ), 2 days a week for 8 weeks, in total 16 sessions.
  Arms: PNF Exercise
Other: Experimental: CTAR Exercise — In addition to the practices in the control group, CTAR exercises will be applied in the presence of a physiotherapist, 2 days a week for 8 weeks, a total of 16 sessions. In the CTAR exercise, the patient is asked to flexion and extension the neck by pressing a standard size and inflatable rubber ball placed under his chin against his sternum. Patients will be asked to do the exercise protocol, which consists of isometric and isotonic components.
  Arms: CTAR Exercise

SUMMARY:
The aim of this study is to examine the effects of PNF (proprioceptive neuromuscular facilitation) and CTAR (Chin Tuck Against Resistance) exercises on swallowing rehabilitation in stroke patients. In addition another aim is to examine the effects of these exercises on the swallowing function, quality of life, functional independence and functional oral intake of individuals, and to investigate the superiority of the exercises to each other in line with these features.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* Who have been diagnosed with stroke
* At least one month has passed since the diagnosis of stroke
* Voluntarily participated in the research,
* Cooperative, able to take instructions (Mini Mental Test score of 24 and above) and
* Individuals with a score of 2 or higher on the Penetration Aspiration Scale will be included.

Exclusion Criteria:

* Lack of long-term sitting balance, unable to maintain an upright position with or without support,
* Have tumors or neoplastic disease in the head and neck region,
* Radiotherapy applied to the neck, swallowing disorders caused by radiotherapy applied to the head and neck region,
* With additional musculoskeletal disease that may cause swallowing disorders,
* With non-stroke neurological disease (Traumatic Brain Injury, Parkinson's, Dementia, ALS, MS, etc.),
* Individuals who have previously received dysphagia treatment will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Penetration Aspiration Scale (PAS) | Change from baseline at 8 weeks
  The penetration aspiration scale (PAS) is routinely used to assess penetration and aspiration severity during videofluoroscopic or FEES assessment. It has a scoring system from 0 to 8, depending on whether it is aspirated or penetrated after administration of liquid-consistent and solid foods with oral contrast agent or dye. High scores indicate the presence of aspiration and penetration.
Ultrasound Evaluation | Change from baseline at 8 weeks
  Neck submental muscle cross-sectional thickness measurement (millimeter-mm), sternocleidomastoideus muscle thickness measurement (mm), hyoid bone elevation measurement (millimeter-mm) and tongue base cross-sectional area (square-centimeter-cm2) will be measured by USG before and after therapy. USG measurements will be made by an experienced radiologist. Three measurements will be taken from each muscle group and the results will be averaged to minimize variations in muscle thickness.

SECONDARY OUTCOMES:
Cognitive Status | a day before the start of treatment
  Mini Mental Test will be used to evaluate the cognitive status of individuals. It is a short, useful, standardized test that provides the opportunity to evaluate cognitive performance in a short time. A high score indicates a good cognitive status. The maximum possible score is 30. A score of 17 and below is considered severe dementia, a score of 18-23 is considered mild dementia, and a score of 24-30 is considered normal.
The Barthel Index | Change from baseline at 8 weeks
  The Barthel index evaluates physical independence in activities of daily living in 10 items (transfer, ambulation/wheelchair use, stair climbing, feeding, dressing, self-regulation, bathing, toilet use, urinary continence, stool continence). Each item is scored separately as 0, 5, 10 or 15 points. A total score of 0-20 means fully dependent, 21-61 highly dependent, 62-90 moderately dependent, 91-99 mildly dependent and 100 fully independent.
Eating Assessment Tool (EAT-10) | Change from baseline at 8 weeks
  It is an easy-to-apply scale consisting of ten items, which allows the rapid assessment of dysphagia symptoms in patients with swallowing disorders. It contains ten questions about oropharyngeal dysphagia, each question is scored between 0 and 3. The total score is obtained by summing the scores. High scores indicate severe dysphagia.
Functional Oral Intake Scale (FOIS) | Change from baseline at 8 weeks
  Oral nutritional status of individuals will be evaluated by using The FOIS is a seven-item scale. It is used to show the level of an individual's feeding tube and oral intake. High scores indicate normal oral intake. The maximum score that can be obtained from the scale is 7.
Swallowing Quality Of Life Questionnaire (SWAL-QOL) | Change from baseline at 8 weeks
  Quality of life due to swallowing problem will be evaluated with the Swallowing Quality of Life Questionnaire (SWAL-QOL). SWAL-QOL includes 10 concepts: general load, food choice, eating time, desire to eat, fear of eating, sleep, fatigue, communication, mental health, and social function. A high score indicates good quality of life. Since its creation, the SWAL-QOL questionnaire has been used as the gold standard in the assessment of quality of life in studies on swallowing disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Nur ÖZCAN, MSc, Principal Investigator — Karamanoğlu Mehmetbey University; Nezehat Özgül ÜNLÜER, PhD, Study Chair — Ankara Yildirim Beyazıt University
Locations (1):
- Selcuk University, Faculty of Medicine, Department of Otolaryngology, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozcan EN, Unluer NO, Ozturk M, Erdur O. Does Proprioceptive Neuromuscular Facilitation Approach Have an Effect on Swallowing Function, Muscle Morphology and Quality of Life in Dysphagic Stroke Patients? A Randomised Controlled Trial. J Oral Rehabil. 2025 Nov;52(11):2044-2058. doi: 10.1111/joor.70000. Epub 2025 Jul 1. PMID 40596755